CLINICAL TRIAL: NCT02739711
Title: Prospective RandomizEd Study Comparing Glycoprotein IIb/IIIa Inhibitors VERsus Standard Therapy in PatientS with Myocardial Infarction and Angiographic Evidence of No-reFLOW
Brief Title: Glycoprotein IIb/IIIa Inhibitors Versus Standard Therapy in Patients with Myocardial Infarction and No-reflow
Acronym: REVERSE-FLOW
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ingo Eitel, Director, Department of Cardiology/Angiology/Intensive Care Medicine, University Heart Center Luebeck, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZ 15-259
Record Dates: First submitted 2016-04-13; First posted 2016-04-15 (Estimated); Last update posted 2025-01-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glycoprotein IIb/IIIa inhibitor (Active Comparator): Glycoprotein IIb/IIIa inhibitor administration
  Interventions: Drug: Glycoprotein IIb/IIIa inhibitors
- Standard therapy (No Intervention): No glycoprotein IIb/IIIa inhibitors

INTERVENTIONS:
Drug: Glycoprotein IIb/IIIa inhibitors — Glycoprotein IIb/IIIa inhibitors intravenous bolus followed by an intravenous infusion for 12/18 h plus medical standard therapy
  Arms: Glycoprotein IIb/IIIa inhibitor

SUMMARY:
Aim of the study is to examine the effects of glycoprotein IIb/IIIa inhibitors on reperfusion success assessed by cardiac magnetic resonance imaging in patients with myocardial infarction and angiographic evidence of no-reflow.

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation myocardial infarction and non-ST-elevation myocardial infarction <48 h after symptom onset
* Angiographic evidence of no-reflow (Thrombolysis in Myocardial Infarction-flow grade ≤2) after primary percutaneous coronary intervention
* Age ≥18 years
* Informed consent

Exclusion Criteria:

* ST-elevation myocardial infarction and non-ST-elevation myocardial infarction patients with Thrombolysis in Myocardial Infarction-flow 3 after primary percutaneous coronary intervention
* Age ≤18 years
* Known pregnancy, breast-feeding or intend to become pregnant during the study period
* Contraindication for treatment with platelet inhibitors
* Known allergy to glycoprotein IIb/IIIa inhibitors, aspirin, or heparin
* Active peptic gastric or duodenal ulcer
* History of major surgery (including intracranial or intraspinal) <4 weeks
* Active bleeding or bleeding diathesis
* Stroke <2 years (ischemic and hemorrhagic)
* Known coagulation defect or relevant thrombocytopenia
* Arteriovenous malformations or aneurysm
* Severe liver insufficiency
* Renal insufficiency requiring dialysis
* Uncontrolled hypertension
* Hypertensive retinopathy
* Vasculitis
* Fibrinolysis <12 hours
* Contraindication for cardiac magnetic resonance imaging at study entry
* Patients without informed consent
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2024-05 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Infarct size assessed by cardiac magnetic resonance imaging | Day 1-10 after myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- University of Luebeck, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eitel I, Saraei R, Jurczyk D, Fach A, Hambrecht R, Wienbergen H, Frerker C, Schmidt T, Allali A, Joost A, Marquetand C, Kurz T, Haaf P, Fahrni G, Mueller C, Desch S, Thiele H, Stiermaier T. Glycoprotein IIb/IIIa inhibitors in acute myocardial infarction and angiographic microvascular obstruction: the REVERSE-FLOW trial. Eur Heart J. 2024 Dec 16;45(47):5058-5067. doi: 10.1093/eurheartj/ehae587. PMID 39217605